CLINICAL TRIAL: NCT07314177
Title: Comparative Effects of Three Dietary Strategies on Body Composition, Metabolic Markers, and Metabolic Syndrome in Adults With Overweight/Obesity: A Randomized Pilot Trial
Brief Title: Effects of Three Dietary Strategies on Body Composition and Metabolic Health in Adults With Overweight or Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI24/171; CEICA-13/2024-PI24-171 (Other Grant/Funding Number: Jane Mateu Foundation)
Record Dates: First submitted 2025-08-28; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Overweight (BMI > 25); Obesity &Amp; Overweight; Metabolic Syndrome (MetS); Cardiometabolic Risk Factors
Keywords: Randomized controlled trial; Mediterranean diet; Low-carbohydrate diet; High-protein diet; Dietary intervention; Metabolic health
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome | interventions — Diet, Mediterranean; Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Mediterranean Diet (Experimental): Participants assigned to this arm will follow a traditional Mediterranean diet providing approximately 55% of total energy from carbohydrates, 15% from protein, and 30% from fats. The diet emphasizes whole grains, fruits, vegetables, legumes, nuts, olive oil as the primary fat source, moderate fish and poultry intake, and limited consumption of red and processed meats, sweets, and sugary beverages. The prescribed energy intake represents a 20-25% caloric deficit based on individual estimated requirements. Participants receive personalized meal plans, nutritional education, and biweekly follow-up by a registered dietitian.
  Interventions: Other: Mediterranean Diet
- Arm 2: Mediterranean Low-Carbohydrate Diet (Experimental): Participants assigned to this arm will follow a Mediterranean-style diet with a reduced carbohydrate content, providing approximately 40% of total energy from carbohydrates, 25% from protein, and 35% from fats. The diet retains the core principles of the Mediterranean pattern, emphasizing vegetables, fruits, legumes, nuts, fish, and olive oil, while limiting bread, pasta, rice, and other high-carbohydrate foods. Energy intake is individualized to achieve a 20-25% caloric deficit. Participants receive personalized meal plans, nutritional education, and biweekly follow-up by a registered dietitian.
  Interventions: Other: Mediterranean Low-Carbohydrate Diet
- Arm 3: High-Protein Diet (Experimental): Participants assigned to this arm will follow a high-protein diet providing approximately 30% of total energy from carbohydrates, 40% from protein, and 30% from fats. Protein sources include lean meats, poultry, fish, eggs, and low-fat dairy products, combined with vegetables, nuts, and healthy fats such as olive oil. Refined carbohydrates and added sugars are limited. Energy intake is individualized to achieve a 20-25% caloric deficit. Participants receive personalized meal plans, nutritional education, and biweekly follow-up by a registered dietitian.
  Interventions: Other: High-Protein Diet

INTERVENTIONS:
Other: Mediterranean Diet — A traditional Mediterranean diet providing approximately 55% of total energy from carbohydrates, 15% from protein, and 30% from fats. Emphasizes whole grains, vegetables, fruits, legumes, nuts, olive oil, moderate fish and poultry, and limited red meat, processed foods, and added sugars. Energy intake adjusted to achieve a 20-25% caloric deficit.
  Arms: Arm 1: Mediterranean Diet
Other: Mediterranean Low-Carbohydrate Diet — A Mediterranean-style diet with reduced carbohydrate content (40% of total energy from carbohydrates, 25% from protein, and 35% from fats). Retains core Mediterranean foods while limiting bread, pasta, rice, and other high-carb foods. Energy intake adjusted to achieve a 20-25% caloric deficit.
  Arms: Arm 2: Mediterranean Low-Carbohydrate Diet
Other: High-Protein Diet — A high-protein dietary pattern providing approximately 30% of total energy from carbohydrates, 40% from protein, and 30% from fats. Includes lean meats, poultry, fish, eggs, low-fat dairy, vegetables, nuts, and olive oil, with limited refined carbs and added sugars. Energy intake adjusted to achieve a 20-25% caloric deficit.
  Arms: Arm 3: High-Protein Diet

SUMMARY:
This study aims to compare the effects of three dietary interventions-a traditional Mediterranean diet, a Mediterranean low-carbohydrate diet, and a high-protein diet-on body composition, metabolic health markers, and metabolic syndrome remission in adults with overweight or obesity. A total of 45 participants will be randomly assigned to one of the three diets for 12 weeks, with regular follow-up by dietitians. Measurements will include weight, body fat, muscle mass, waist and hip circumference, blood pressure, and blood tests to assess glucose, cholesterol, inflammation, and other metabolic parameters. The findings will help determine whether one dietary pattern is more effective than others in improving short-term health outcomes in this population.

DETAILED DESCRIPTION:
Detailed Description:

This randomized, controlled, parallel-group pilot clinical trial will evaluate the effects of three different hypocaloric dietary strategies on body composition, metabolic markers, and metabolic syndrome remission in adults with overweight or obesity.

Background and Rationale Overweight and obesity are highly prevalent in Europe and are associated with an increased risk of metabolic syndrome, cardiovascular disease, type 2 diabetes, and obesity-related cancers. Dietary interventions are a cornerstone in their management, but the optimal macronutrient composition for improving short-term metabolic outcomes remains unclear. This study investigates the comparative impact of a traditional Mediterranean diet, a Mediterranean low-carbohydrate diet, and a high-protein diet over a 12-week period.

Study Design A total of 45 participants aged 18-65 years with a body mass index (BMI) ≥25 kg/m² will be recruited through online advertisements and primary care referrals. After eligibility screening and informed consent, participants will be randomly allocated (1:1:1) to one of the three dietary intervention arms.

Intervention

All diets will be hypocaloric, aiming for a 20-25% reduction in individual energy requirements, and will differ in macronutrient distribution:

Mediterranean diet: 55% carbohydrates, 15% proteins, 30% fats.

Mediterranean low-carbohydrate diet: 40% carbohydrates, 25% proteins, 35% fats.

High-protein diet: 30% carbohydrates, 40% proteins, 30% fats.

Participants will be followed biweekly by qualified dietitians through in-person or phone consultations. They will receive personalized meal plans, nutritional education, and support materials to enhance adherence.

Assessments Anthropometric measures (BMI, fat mass, fat-free mass, waist and hip circumference) will be obtained at baseline and at 12 weeks using standardized protocols and validated equipment. Blood pressure will be measured with a calibrated automated device after a seated rest. Fasting blood samples will be collected in the morning for biochemical analyses, including glucose, HbA1c, insulin, lipid profile, uric acid, iron status, high-sensitivity C-reactive protein, fibrinogen, erythrocyte sedimentation rate, and liver enzymes.

Outcomes The primary outcome is the change in BMI after 12 weeks. Secondary outcomes include changes in body composition, metabolic and inflammatory biomarkers, and the proportion of participants meeting the International Diabetes Federation (IDF) criteria for metabolic syndrome at baseline and post-intervention.

Ethics and Dissemination The study protocol was approved by the Ethics Committee of Aragón (CEICA) (No. 13/2024) and will be conducted in accordance with the Declaration of Helsinki and current regulatory requirements. The findings will be disseminated through peer-reviewed publications and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-70 years
* Body mass index (BMI) ≥ 25 kg/m² (overweight or obesity)
* Stable body weight (± 2 kg) in the last 3 months prior to screening
* Willingness to follow one of the prescribed dietary interventions for 12 weeks
* Ability to attend scheduled follow-up visits and complete study assessments
* Provided written informed consent prior to study participation

Exclusion Criteria:

* Diagnosis of type 1 diabetes, cardiovascular disease, cancer, chronic kidney disease, liver disease, or other serious chronic conditions that could interfere with the intervention
* Pregnancy or breastfeeding
* Current participation in another clinical trial
* History of bariatric surgery or weight-loss program within the past 6 months
* Use of medications known to affect body weight, metabolism, or appetite (e.g., glucocorticoids, weight-loss drugs, antipsychotics)
* Any food allergy or intolerance that would preclude adherence to the assigned diet
* Alcohol or substance abuse
* Any condition or circumstance that, in the opinion of the investigators, would make the participant unsuitable for the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-09-08 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI, kg/m²) assessed by weight (Tanita MC-780MA bioimpedance scale) and height (Seca stadiometer) from baseline to 12 weeks | Baseline and week 12
  BMI will be calculated as weight (kg) divided by height (m²). Weight will be measured without shoes using a Tanita MC-780MA multi-frequency bioelectrical impedance analyzer, and height will be measured using a calibrated Seca wall-mounted stadiometer.

SECONDARY OUTCOMES:
Change in Fat Mass Percentage (%) assessed by Tanita MC-780MA bioelectrical impedance analyzer from baseline to 12 weeks | Baseline and week 12
  Fat mass percentage will be estimated using multi-frequency segmental bioelectrical impedance analysis (Tanita MC-780MA).
Change in Fat-Free Mass Percentage (%) assessed by Tanita MC-780MA bioelectrical impedance analyzer from baseline to 12 weeks | Baseline and week 12
  Fat-free mass percentage will be estimated using multi-frequency segmental bioelectrical impedance analysis (Tanita MC-780MA).
Change in Metabolic Syndrome Status (yes/no) defined by IDF criteria from baseline to 12 weeks | Baseline and week 12
  Metabolic syndrome will be diagnosed according to the International Diabetes Federation (IDF) criteria, requiring ≥3 of the following: elevated waist circumference, elevated triglycerides, reduced HDL cholesterol, elevated blood pressure, or elevated fasting glucose.
Change in glycated hemoglobin (HbA1c, %) from baseline to 12 weeks | Baseline and week 12
  HbA1c levels will be measured in fasting venous blood samples using high-performance liquid chromatography (HPLC), following standardized laboratory procedures.
Change in serum total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides (mg/dL) from baseline to 12 weeks | Baseline and week 12
  Serum lipids will be determined from fasting blood samples analyzed enzymatically in a certified laboratory. Results will be reported in mg/dL for each parameter.
Change in fasting glucose (mg/dL) from baseline to 12 weeks | Baseline and week 12
  Fasting glucose concentration will be measured in venous blood samples collected early in the morning under standardized fasting conditions. Glucose levels will be quantified using validated automated enzymatic assays in a certified clinical laboratory.
Change in high-sensitivity C-reactive protein (hs-CRP, mg/dL) from baseline to 12 weeks | Baseline and week 12
  Serum hs-CRP concentrations will be measured in fasting venous blood samples collected in the morning and analyzed using a standardized high-sensitivity immunoassay in a certified clinical laboratory. Values will be reported in mg/dL.
Change in serum uric acid (mg/dL) from baseline to 12 weeks | Baseline and week 12
  Serum uric acid will be measured by an enzymatic colorimetric method in a certified laboratory. Results will be reported in mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Edificio SAI, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No